CLINICAL TRIAL: NCT01168973
Title: A Randomized, Double-Blind, Phase 3 Study of Docetaxel and Ramucirumab Versus Docetaxel and Placebo in the Treatment of Stage IV Non-Small Cell Lung Cancer Following Disease Progression After One Prior Platinum-Based Therapy
Brief Title: A Study of Chemotherapy and Ramucirumab Versus Chemotherapy Alone in Second Line Non-Small Cell Lung Cancer (NSCLC) Participants Who Received Prior First Line Platinum-based Chemotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13852; I4T-MC-JVBA (Other: Eli Lilly and Company); 2010-021297-11 (EudraCT Number); CP12-1027 (Other: ImClone Trial Number); CTRI/2011/08/001942 (Registry Identifier: Clinical Trials Registry India)
Record Dates: First submitted 2010-07-16; First posted 2010-07-23 (Estimated); Results first posted 2014-12-29 (Estimated); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: second line; non small cell lung cancer; NSCLC; phase 3; ramucirumab; lung cancer; docetaxel; taxotere
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Ramucirumab; Docetaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ramucirumab + Docetaxel (Experimental)
  Interventions: Biological: Ramucirumab; Drug: Docetaxel
- Placebo + Docetaxel (Placebo Comparator)
  Interventions: Drug: Placebo (for Ramucirumab); Drug: Docetaxel

INTERVENTIONS:
Biological: Ramucirumab — 10 milligrams per kilogram (mg/kg) administered intravenously (IV) on Day 1 of 21-day cycle until disease progression, unacceptable toxicity, or another withdrawal criterion is met
  Other Names: IMC 1121B; LY3009806
  Arms: Ramucirumab + Docetaxel
Drug: Placebo (for Ramucirumab) — Administered IV on Day 1 of 21-day cycle until disease progression, unacceptable toxicity, or another withdrawal criterion is met
  Arms: Placebo + Docetaxel
Drug: Docetaxel — 75 milligrams per square meter (mg/m^2) (60 mg/m^2 for the countries of Korea and Taiwan only with protocol amendment dated 22 May 2012) administered IV on Day 1 of 21-day cycle until disease progression, unacceptable toxicity, or another withdrawal criterion is met

SUMMARY:
The purpose of the study is to compare the survival of participants who receive chemotherapy and ramucirumab versus chemotherapy alone as second line treatment for NSCLC after prior first line platinum-based chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Disease progression during or after one prior first-line platinum-based chemotherapy with or without maintenance therapy
* Prior bevacizumab as first-line and/or maintenance therapy is allowed
* Signed informed consent
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Histologically or cytologically confirmed NSCLC
* Stage IV NSCLC disease
* Participants have measurable or nonmeasurable disease
* Adequate organ function, defined as:

  * Total bilirubin less than or equal to Upper Limit of Normal (ULN),
  * Aspartate Aminotransferase (AST) and Alanine Aminotransaminase (ALT) less than or equal to 2.5 x ULN, or less than or equal to 5 x ULN if the transferase elevation is due to liver metastases,
  * Serum creatinine less than or equal to 1.5 x ULN or calculated creatinine clearance greater than or equal to 50 milliliters per minute (ml/min) (per the Cockcroft-Gault formula or equivalent and/or 24-hour urine collection),
  * Absolute Neutrophil Count (ANC) greater than or equal to 1.5 x 10^3/microliters (µL), hemoglobin greater than or equal to 10.0 grams/deciliter (g/dL), and platelets greater than or equal to 100 x 10^3/µL,
  * Adequate coagulation function as defined by International Normalized Ratio (INR) less than or equal to 1.5, or prothrombin time and partial thromboplastin time less than or equal to 1.5 x ULN.
  * The participant does not have cirrhosis at a level of Child-Pugh B (or worse) or cirrhosis (any degree) and a history of hepatic encephalopathy or clinically meaningful ascites resulting from cirrhosis. Clinically meaningful ascites is defined as ascites resulting from cirrhosis and requiring ongoing treatment with diuretics and/or paracentesis.
* Urinary protein is less than or equal to 1+ on dipstick or routine urinalysis. If urine dipstick or routine analysis indicates proteinuria greater than or equal to 2+, a 24-hour urine must be collected and must demonstrate less than 1000 milligrams (mg) of protein.
* Participants of reproductive potential (both sexes) must agree to use reliable method of birth control (hormonal or barrier methods) during the study period and at least 12 weeks after the last dose of study therapy
* Life expectancy of greater than or equal to 3 months
* Prior radiation therapy is allowed if: In the case of chest radiotherapy at least 28 days have elapsed from the completion of radiation treatment prior to randomization; In the case of focal or palliative radiation treatment at least 7 days have elapsed from last radiation treatment prior to randomization (and provided that 25% or less of total bone marrow had been irradiated); In the case of Central Nervous System (CNS) radiation at least 14 days have elapsed from the completion of radiation treatment prior to randomization

Exclusion Criteria:

* Disease progression on more than 1 prior chemotherapy regimens
* Participants whose only prior treatment was a tyrosine kinase inhibitor
* The participant's tumor wholly or partially contains small cell lung cancer
* Major surgery within 28 days prior to randomization, or subcutaneous venous access device placement within 7 days prior to randomization. Postoperative bleeding complications or wound complications from a surgical procedure performed in the last 2 months.
* Concurrent treatment with other anticancer therapy, including other chemotherapy, immunotherapy, hormonal therapy, chemoembolization, or targeted therapy
* Last dose of bevacizumab must be at least 28 days from time of randomization
* Last dose of cytotoxic chemotherapy must be at least 14 days from time of randomization
* The participant has untreated CNS metastases. Participants with treated brain metastases are eligible if they are clinically stable with regard to neurologic function, off steroids after cranial irradiation ending at least 2 weeks prior to randomization, or after surgical resection performed at least 28 days prior to randomization. No evidence of Grade greater than or equal to 1 CNS hemorrhage based on pretreatment Magnetic Resonance Imaging (MRI) or IV contrast Computed Tomography (CT) scan.
* Radiologically documented evidence of major blood vessel invasion or encasement by cancer
* Radiographic evidence of intratumor cavitation
* History of uncontrolled hereditary or acquired thrombotic disorder
* Chronic therapy with nonsteroidal anti-inflammatory drug (NSAIDs) or other antiplatelet agents; Aspirin use at doses up to 325 milligrams per day (mg/day) is permitted
* History of gross hemoptysis (defined as bright red blood or greater than or equal to 1/2 teaspoon) within 2 months prior to randomization
* Clinically relevant congestive heart failure [New York Heart Association (NYHA II-IV)] or symptomatic or poorly controlled cardiac arrhythmia
* Any arterial thrombotic event, including myocardial infarction, unstable angina, cerebrovascular accident, or transient ischemic attack, within 6 months prior to randomization
* Uncontrolled arterial hypertension greater than or equal to 150 / greater than or equal to 90 millimeters of mercury (mm Hg) despite standard medical management
* Serious or nonhealing wound, ulcer, or bone fracture within 28 days prior to randomization
* Significant bleeding disorders, vasculitis, or Grade 3/4 gastrointestinal bleeding within 3 months prior to randomization
* Gastrointestinal (GI) perforation and/or fistulae within 6 months prior to randomization
* Bowel obstruction, history or presence of inflammatory enteropathy or extensive intestinal resection Crohn's disease, ulcerative colitis, or chronic diarrhea
* Peripheral neuropathy greater than or equal to Grade 2 [National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 4.02]
* Serious illness or medical condition(s) including, but not limited to: Human immunodeficiency virus (HIV) infection or acquired immunodeficiency syndrome (AIDS)-related illness; Active or uncontrolled clinically serious infection; Severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration
* Known allergy or hypersensitivity reaction to any of the treatment components
* The participant is pregnant or breastfeeding
* Current or recent (within 28 days prior to randomization) treatment with an investigational drug or device that has not received regulatory approval for any indication at the time of randomization, or participation in another interventional clinical trial
* Prior therapy with docetaxel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1253 (Actual)
Dates: Start 2010-12; Primary Completion 2013-12 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9AM - 5PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (230):
- United States (96):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Phoenix, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sedona, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fayetteville, Arkansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Alhambra, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Duarte, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fresno, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fullerton, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., La Jolla, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Long Beach, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Los Angeles, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Northridge, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Redondo Beach, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santa Barbara, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santa Monica, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Denver, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Waterbury, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jacksonville, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Miami, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ocala, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orlando, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Athens, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Augusta, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lawrenceville, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Macon, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rome, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Savannah, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Springfield, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bloomington, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cedar Rapids, Iowa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Iowa City, Iowa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Overland Park, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wichita, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ashland, Kentucky
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mount Sterling, Kentucky
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Baton Rouge, Louisiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Metairie, Louisiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bethesda, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chevy Chase, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Boston, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Danvers, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Framingham, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Newton, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ann Arbor, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Minneapolis, Minnesota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Columbia, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Joplin, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St Louis, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Billings, Montana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Henderson, Nevada
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Reno, Nevada
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lebanon, New Hampshire
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Portsmouth, New Hampshire
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Albuquerque, New Mexico
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Latham, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New York, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., The Bronx, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Durham, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Raleigh, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fargo, North Dakota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Columbus, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tulsa, Oklahoma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Abington, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kingston, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Philadelphia, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Charleston, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sioux Falls, South Dakota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chattanooga, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Memphis, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Abilene, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Amarillo, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beaumont, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bedford, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., El Paso, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fort Worth, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lewisville, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., McAllen, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mesquite, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Midland, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Odessa, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Paris, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Antonio, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sherman, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sugar Land, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., The Woodlands, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tyler, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Webster, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wichita Falls, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Christiansburg, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fairfax, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Newport News, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Richmond, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lacey, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Spokane, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wenatchee, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madison, Wisconsin
- Argentina (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Buenos Aires
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Córdoba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., La Rioja
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rosario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tucumain
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Viedma
- Austria (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Graz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Grimmenstein
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vienna
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wels
- Brazil (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barretos
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Belo Horizonte
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Goiânia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Porto Alegre
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., São Paulo
- Canada (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Edmonton, Alberta
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Moncton, New Brunswick
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sainte-Foy, Quebec
- France (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Grenoble
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lille
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lyon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nice
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Strasbourg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toulouse
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vandœuvre-lès-Nancy
- Germany (13):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Augsburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bad Soden
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bielefeld
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dresden
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Frankfurt
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gerlingen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Großhansdorf
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Halle
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Heidelberg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Immenhausen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oldenburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ulm
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Villingen-Schwenningen
- Greece (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Athens
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kifissia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pátrai
- Hungary (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Budapest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gyula
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mátraháza
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nyíregyháza
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pécs
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Székesfehérvár
- India (9):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bangalore
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cuttack
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Delhi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jaipur
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kochi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madurai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mumbai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pune
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Trivandrum
- Israel (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Haifa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jerusalem
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kfar Saba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Petah Tikva
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Safed
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tel Aviv
- Italy (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Livorno
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Monza
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Novara
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Padua
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Palermo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Parma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pisa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rome
- Mexico (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guadalajara
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mexico City
- Netherlands (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., 's-Hertogenbosch
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Amsterdam
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Arnhem
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Harderwijk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zwolle
- New Zealand (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Grafton
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wellington
- Norway (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oslo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tromsø
- Poland (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gdansk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gdynia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Głuchołazy
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Krakow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lodz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Opole
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Otwock
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Poznan
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bayamón, Puerto Rico
- Romania (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bucharest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cluj-Napoca
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Iași
- Russia (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Moscow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint Petersburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Stavropol
- South Korea (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Incheon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seoul
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Suwon
- Spain (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Girona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Las Palmas de Gran Canaria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madrid
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mataró
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pamplona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pozuelo de Alarcón
- Sweden (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Eskilstuna
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Linköping
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lund
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Solna
- Switzerland (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Basel
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bern
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fribourg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lucerne
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zurich
- Taiwan (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kaohsiung City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kuei Shan Hsiang
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Neihu Taipei
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Niao Sung Hsiang
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taichung
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taipei
- Turkey (Türkiye) (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ankara
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Istanbul
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Izmir
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kayseri
- United Kingdom (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cottingham, East Yorkshire
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., London, Greater London
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Preston, Lancashire
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wythenshawe, Manchester
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Scunthorpe, North Lincolnshire
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Glasgow, Scotland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Coventry, West Midlands
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wolverhampton, West Midlands

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Rolfo C, Hess LM, Jen MH, Peterson P, Li X, Liu H, Lai Y, Sugihara T, Kiiskinen U, Vickers A, Summers Y. External control cohorts for the single-arm LIBRETTO-001 trial of selpercatinib in RET+ non-small-cell lung cancer. ESMO Open. 2022 Aug;7(4):100551. doi: 10.1016/j.esmoop.2022.100551. Epub 2022 Aug 2. PMID 35930972
- [Derived] Garon EB, Scagliotti GV, Gautschi O, Reck M, Thomas M, Iglesias Docampo L, Kalofonos H, Kim JH, Gans S, Brustugun OT, Orlov SV, Cuyun Carter G, Zimmermann AH, Oton AB, Alexandris E, Lee P, Wolff K, Stefaniak VJ, Socinski MA, Perol M. Exploratory analysis of front-line therapies in REVEL: a randomised phase 3 study of ramucirumab plus docetaxel versus docetaxel for the treatment of stage IV non-small-cell lung cancer after disease progression on platinum-based therapy. ESMO Open. 2020 Jan;5(1):e000567. doi: 10.1136/esmoopen-2019-000567. PMID 31958290
- [Derived] Garon EB, Ciuleanu TE, Arrieta O, Prabhash K, Syrigos KN, Goksel T, Park K, Gorbunova V, Kowalyszyn RD, Pikiel J, Czyzewicz G, Orlov SV, Lewanski CR, Thomas M, Bidoli P, Dakhil S, Gans S, Kim JH, Grigorescu A, Karaseva N, Reck M, Cappuzzo F, Alexandris E, Sashegyi A, Yurasov S, Perol M. Ramucirumab plus docetaxel versus placebo plus docetaxel for second-line treatment of stage IV non-small-cell lung cancer after disease progression on platinum-based therapy (REVEL): a multicentre, double-blind, randomised phase 3 trial. Lancet. 2014 Aug 23;384(9944):665-73. doi: 10.1016/S0140-6736(14)60845-X. Epub 2014 Jun 2. PMID 24933332
- [Derived] Garon EB, Cao D, Alexandris E, John WJ, Yurasov S, Perol M. A randomized, double-blind, phase III study of Docetaxel and Ramucirumab versus Docetaxel and placebo in the treatment of stage IV non-small-cell lung cancer after disease progression after 1 previous platinum-based therapy (REVEL): treatment rationale and study design. Clin Lung Cancer. 2012 Nov;13(6):505-9. doi: 10.1016/j.cllc.2012.06.007. Epub 2012 Jul 31. PMID 22853980

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who died, due to any cause, or were alive at the end of the study but off study drug were considered to have completed the study.
Groups:
- Ramucirumab and Docetaxel: On Day 1 of each 21-day cycle, participants received ramucirumab drug product (DP) followed by docetaxel. Treatment continued until disease progression, unacceptable toxicity, or other withdrawal criteria were met.
  * Ramucirumab DP: 10 milligrams per kilogram (mg/kg) administered intravenously.
  * Docetaxel: 75 milligrams per square meter (mg/m^2) (60 mg/m^2 for the countries of Korea and Taiwan only, with protocol amendment dated 22 May 2012) administered intravenously.
- Placebo and Docetaxel: On Day 1 of each 21-day cycle, participants received placebo followed by docetaxel. Treatment continued until disease progression, unacceptable toxicity, or other withdrawal criteria were met.
  * Placebo (matching Ramucirumab DP): 10 mg/kg administered intravenously.
  * Docetaxel: 75 mg/m^2 (60 mg/m^2 for the countries of Korea and Taiwan only, with protocol amendment dated 22 May 2012) administered intravenously.
Period: Overall Study
Arm/Group | Ramucirumab and Docetaxel | Placebo and Docetaxel
Started | 628 | 625
Received Any Quantity of Any Study Drug | 624 | 621 (Three participants randomized to placebo and docetaxel received 1 dose of ramucirumab in error.)
Completed | 15 | 14
Not Completed | 613 | 611
Not completed — Progressive Disease | 341 | 429
Not completed — Adverse Event | 94 | 55
Not completed — Withdrawal by Subject | 90 | 53
Not completed — Death | 42 | 45
Not completed — Physician Decision | 37 | 19
Not completed — Sponsor Decision | 2 | 1
Not completed — Protocol Criterion Not Met and Deviation | 7 | 9

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) population: All randomized participants grouped according to their assigned treatment at randomization.
Groups:
- Ramucirumab and Docetaxel: On Day 1 of each 21-day cycle, participants received ramucirumab DP followed by docetaxel. Treatment continued until disease progression, unacceptable toxicity, or other withdrawal criteria were met.
  * Ramucirumab DP: 10 mg/kg administered intravenously.
  * Docetaxel: 75 mg/m^2 (60 mg/m^2 for the countries of Korea and Taiwan only, with protocol amendment dated 22 May 2012) administered intravenously.
- Total: Total of all reporting groups
Arm/Group | Ramucirumab and Docetaxel | Placebo and Docetaxel | Total
Number analyzed (Participants) | 628 | 625 | 1253
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 391 | 407 | 798
  >=65 years | 237 | 218 | 455
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 209 | 210 | 419
  Male | 419 | 415 | 834
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 43 | 53 | 96
  Not Hispanic or Latino | 387 | 380 | 767
  Unknown or Not Reported | 198 | 192 | 390
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 9 | 20 | 29
  Asian | 74 | 86 | 160
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 17 | 16 | 33
  White | 526 | 503 | 1029
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 156 | 152 | 308
  Taiwan | 9 | 18 | 27
  Greece | 25 | 19 | 44
  Spain | 27 | 23 | 50
  Israel | 14 | 8 | 22
  Russian Federation | 28 | 33 | 61
  Italy | 26 | 28 | 54
  Switzerland | 12 | 14 | 26
  India | 22 | 33 | 55
  France | 21 | 24 | 45
  Puerto Rico | 1 | 2 | 3
  Netherlands | 15 | 16 | 31
  Korea, Republic of | 34 | 28 | 62
  Turkey | 22 | 23 | 45
  Austria | 11 | 9 | 20
  United Kingdom | 19 | 19 | 38
  Hungary | 9 | 4 | 13
  Mexico | 11 | 20 | 31
  Canada | 12 | 7 | 19
  Argentina | 16 | 17 | 33
  Brazil | 4 | 3 | 7
  Poland | 30 | 33 | 63
  Romania | 41 | 36 | 77
  Norway | 10 | 3 | 13
  Germany | 40 | 42 | 82
  New Zealand | 3 | 4 | 7
  Sweden | 10 | 7 | 17

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Overall survival was the time from randomization until the date of death from any cause. Participants who were alive at the end of the follow-up period (or lost to follow-up) were censored on the last date the participant was known to be alive.
Time Frame: Randomization to date of death from any cause (up to 34 months)
Population: Intent-to-Treat (ITT) population: All randomized participants grouped according to their assigned treatment at randomization. Participants censored: ramucirumab and docetaxel arm = 200 participants; placebo and docetaxel arm = 169 participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ramucirumab and Docetaxel | Placebo and Docetaxel
Number analyzed (Participants) | 628 | 625
months | 10.5 [9.5 to 11.2] | 9.1 [8.4 to 10.0]

2. Secondary Outcome: Progression-Free Survival (PFS) Time
Description: PFS time was the time from randomization until the date of objectively determined progressive disease (PD) or death due to any cause, whichever occurred first. According to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1), PD was at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study. In addition to the 20% relative increase, the sum must have also demonstrated an absolute increase of at least 5 millimeters (mm). The appearance of 1 or more new lesions and/or unequivocal progression of existing nontarget lesions was also considered progression. Participants without objectively determined PD who were alive at the end of the follow-up period (or lost to follow-up) were censored on the date of the participant's last complete radiographic tumor assessment; if no baseline or post-baseline radiologic assessment was available, the participant was censored at the date of randomization.
Time Frame: Randomization to measured PD or date of death from any cause (up to 29 months)
Population: ITT population: All randomized participants grouped according to their assigned treatment at randomization. Participants censored: ramucirumab and docetaxel arm = 70 participants; placebo and docetaxel arm = 42 participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ramucirumab and Docetaxel | Placebo and Docetaxel
Number analyzed (Participants) | 628 | 625
months | 4.5 [4.2 to 5.3] | 3.0 [2.8 to 3.9]

3. Secondary Outcome: Percentage of Participants Achieving an Objective Response (Objective Response Rate)
Description: Participants achieved an objective response if they had a best overall response of partial response (PR) or complete response (CR). According to RECIST v1.1, PR was defined as at least a 30% decrease in the sum of the diameters of target lesions (including the short axes of any target lymph node), taking as reference the baseline sum diameter; CR was the disappearance of all non-nodal target lesions, with the short axes of any target lymph node reduced to <10 mm, the disappearance of all nontarget lesions, and the normalization of tumor marker levels [if tumor markers were initially above the upper limit of normal (ULN)]. The percentage of participants who achieved an objective response=(number of participants with CR or PR)/(number of participants assessed)*100.
Time Frame: Baseline to measured PD (up to 29 months)
Population: ITT population: All randomized participants grouped according to their assigned treatment at randomization.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ramucirumab and Docetaxel | Placebo and Docetaxel
Number analyzed (Participants) | 628 | 625
percentage of participants | 22.9 [19.7 to 26.4] | 13.6 [11.0 to 16.5]

4. Secondary Outcome: Percentage of Participants Achieving Disease Control (Disease Control Rate)
Description: Participants achieved disease control if they had a best overall response of PR, CR or stable disease (SD). According to RECIST v1.1, PR was defined as at least a 30% decrease in the sum of the diameters of target lesions (including the short axes of any target lymph node), taking as reference the baseline sum diameter; CR was the disappearance of all non-nodal target lesions, with the short axes of any target lymph node reduced to <10 mm, the disappearance of all nontarget lesions, and the normalization of tumor marker levels (if tumor markers were initially above the ULN). SD was neither sufficient shrinkage to qualify as PR nor sufficient increase to qualify as PD, taking as reference the smallest sum diameter since treatment started. The percentage of participants who achieved disease control=(number of participants with CR, PR, or SD)/(number of participants assessed)*100.
Time Frame: Baseline to measured PD (up to 29 months)
Population: ITT population: All randomized participants grouped according to their assigned treatment at randomization.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ramucirumab and Docetaxel | Placebo and Docetaxel
Number analyzed (Participants) | 628 | 625
percentage of participants | 64.0 [60.1 to 67.8] | 52.6 [48.6 to 56.6]

5. Secondary Outcome: Maximum Improvement on Lung Cancer Symptom Scale (LCSS)
Description: The LCSS consisted of 9 items: 6 items focused on lung cancer symptoms [loss of appetite, fatigue, cough, dyspnea (shortness of breath), hemoptysis (blood in sputum), and pain] and 3 items were global items (symptom distress, interference with activity level, and global quality of life). Participant responses to each item were measured using visual analogue scales (VAS) with 100-mm lines. A higher score for any item represented a higher level of symptoms/problems. The Average Symptom Burden Index (ASBI) was the mean of the 6 symptom items of the LCSS, and the Total LCSS was the mean of all 9 LCSS items. ASBI and Total LCSS were not computed for a participant if he/she had 1 or more missing values for the 6 and 9 items, respectively. Maximum improvement in LCSS scores, ASBI, and Total LCSS score was the largest decrease from baseline for each variable, which was the smallest (most negative or smallest positive) non-missing value among all change from baseline values for each variable.
Time Frame: Baseline, Day 21 of each cycle, and 30 days following last infusion (up to Cycle 38, 21 days/cycle)
Population: Randomized participants grouped according to their assigned treatment at randomization, who had a baseline and at least 1 post-baseline LCSS score.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Ramucirumab and Docetaxel | Placebo and Docetaxel
Number analyzed (Participants) | 476 | 477
mm
  Loss of Appetite (n=473, 471) | -10.9 (26.11) | -11.0 (26.22)
  Fatigue (n=473, 472) | -12.1 (23.86) | -12.0 (27.29)
  Cough (n=476, 473) | -13.8 (24.28) | -14.3 (26.28)
  Dyspnea (n=472, 477) | -11.0 (23.01) | -10.5 (24.31)
  Hemoptysis (n=475, 475) | -1.4 (8.89) | -1.1 (8.79)
  Pain (n=476, 475) | -11.3 (23.62) | -11.5 (24.85)
  Symptom Distress (n=474, 472) | -10.7 (23.37) | -12.2 (26.25)
  Interference With Activity Level (n=474, 472) | -8.5 (24.13) | -7.9 (24.95)
  Global Quality of Life (n=467, 469) | -10.4 (22.68) | -8.9 (23.23)
  ASBI (n=455, 456) | -6.1 (13.75) | -6.9 (14.50)
  Total LCSS (n=446, 446) | -5.2 (13.75) | -6.4 (14.66)

6. Secondary Outcome: Change From Baseline to 30-Day Follow-Up Visit on European Quality of Life Questionnaire-5 Dimension (EQ-5D) Health State Scores
Description: The EQ-5D is a quality-of-life instrument that consists of 2 parts. The first part (Health State Index score) allowed participants to rate their health state in 5 health domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression using a scale from 1 to 3 (no problem, some problems, and extreme problems, respectively). These combinations of attributes were converted into a weighted Health State Index score according to a United Kingdom population-based algorithm; the possible values for the Health State Index score ranged from -0.59 (severe problems in all 5 dimensions) to 1.0 (no problem in any dimension). The second part of the EQ-5D was a VAS that allowed participants to rate their present health condition. Possible EQ-5D VAS scores ranged from 0 (worst imaginable health state) to 100 (best imaginable health state).
Time Frame: Baseline, 30 days following last infusion (up to Cycle 38, 21 days/cycle)
Population: Randomized participants grouped according to their assigned treatment at randomization, who had an EQ-5D assessment at a baseline and 30 days post treatment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ramucirumab and Docetaxel | Placebo and Docetaxel
Number analyzed (Participants) | 272 | 272
units on a scale
  Health State Index Score (n=266, 272) | -0.140 (0.308) | -0.126 (0.294)
  Health State VAS Score (n=272, 254) | -5.9 (21.02) | -6.1 (20.31)

7. Secondary Outcome: Maximum and Minimum Serum Concentrations (Cmax and Cmin) of Ramucirumab
Time Frame: Prior to infusion and 1 hour following infusion for 4 and 8 (cycles 3 and 5 at 21 days/cycle)
Population: Participants assigned to the ramucirumab and docetaxel arm at randomization, who had evaluable ramucirumab pharmacokinetic (PK) data to calculate Cmax and Cmin.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (mcg/mL)
Arm/Group | Ramucirumab and Docetaxel
Number analyzed (Participants) | 594
micrograms per milliliter (mcg/mL)
  Cmax at Cycle 3 | 262 (30)
  Cmin at Cycle 3 | 28.3 (65)
  Cmax at Cycle 5 | 237 (38)
  Cmin at Cycle 5 | 38.4 (63)

8. Secondary Outcome: Number of Participants With Anti-Ramucirumab Antibodies
Description: The number of participants who had treatment-emergent or follow-up emergent anti-drug antibodies (ADA) is reported. Participants with treatment-emergent ADA were defined as participants who had any sample from baseline through Cycle 5 pre-infusion that was a 4-fold increase (2 dilution increase) in immunogenicity titer over the baseline titer, or participants who tested negative at baseline and positive post-baseline (at titer of ≥1:20). Participants with follow-up emergent ADA were defined as participants who had any sample during 30 days post last infusion that was a 4-fold increase (2 dilution increase) in immunogenicity titer over the baseline titer.
Time Frame: Baseline, prior to infusion for week 4 and 8 (cycles 3 and 5), and 30 days following last infusion (up to Cycle 38, 21 days/cycle)
Population: Randomized participants who received any quantity of study treatment, grouped by the treatment they actually received, who had a baseline and at least 1 post-baseline ADA assessment.
Measure: Number; unit: participants
Arm/Group | Ramucirumab and Docetaxel | Placebo and Docetaxel
Number analyzed (Participants) | 599 | 598
participants
  Treatment-Emergent ADA (n=599, 598) | 9 | 16
  Follow-Up Emergent ADA (n=506, 481) | 9 | 16

9. Other Pre Specified Outcome: Number of Participants Who Had Treatment-Emergent Adverse Events (TEAEs) or Died
Description: Data presented are the number of participants who experienced at least 1 TEAE, Grade 3, 4, or 5 TEAE, treatment-emergent serious adverse event (SAE), TEAE leading to discontinuation of study treatment (ramucirumab/placebo or docetaxel), and TEAE leading to death. Clinically significant events were defined as treatment-emergent SAEs and other non-serious adverse events (AEs) regardless of causality. A summary of SAEs and other non-serious AEs, regardless of causality, is located in the Reported Adverse Events module.
Time Frame: First infusion up to 30 days following last infusion (up to Cycle 38, 21 days/cycle)
Population: Safety population: Randomized participants who received any quantity of study drug, grouped by the treatment they actually received.
Measure: Number; unit: participants
Arm/Group | Ramucirumab and Docetaxel | Placebo and Docetaxel
Number analyzed (Participants) | 627 | 618
participants
  At least 1 TEAE | 613 | 594
  At least 1 Grade 3, 4, or 5 TEAE | 495 | 444
  At least 1 treatment-emergent SAE | 269 | 262
  TEAE leading to study drug discontinuation | 58 | 32
  TEAE leading to death | 34 | 35
  Deaths While On Treatment | 428 | 451
  Deaths During 30 Days Post Last Dose | 53 | 58

ADVERSE EVENTS:
Time Frame: Randomization through 30 days following last infusion (up to Cycle 38, 21 days/cycle).
Description: Safety Population: All randomized participants who received any quantity of study treatment, grouped by the treatment they actually received.
  Three participants randomized to placebo and docetaxel received 1 dose of ramucirumab in error.
Arm/Group | Ramucirumab and Docetaxel | Placebo and Docetaxel
Serious Adverse Events (participants affected / at risk) | 284/627 | 281/618
Other Adverse Events (participants affected / at risk) | 601/627 | 583/618
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ramucirumab and Docetaxel (N=627) | Placebo and Docetaxel (N=618)
Anaemia (Blood and lymphatic system disorders) | 10 (16) | 14 (17)
Febrile neutropenia (Blood and lymphatic system disorders) | 86 (104) | 51 (56)
Leukopenia (Blood and lymphatic system disorders) | 5 (6) | 10 (14)
Neutropenia (Blood and lymphatic system disorders) | 30 (38) | 27 (33)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 6 (6) | 2 (2)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac arrest (Cardiac disorders) | 2 (2) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 1 (2) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 2 (2) | 2 (2)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (2) | 6 (6)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 2 (2) | 3 (4)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Tracheo-oesophageal fistula (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Diplopia (Eye disorders) | 1 (1) | 0 (0)
Retinal vein thrombosis (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 7 (8)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal inflammation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (2) | 0 (0)
Colitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 13 (13) | 9 (9)
Diverticular perforation (Gastrointestinal disorders) | 2 (2) | 2 (2)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 3 (4)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 2 (3)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gingival bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 2 (2) | 0 (0)
Ileus paralytic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 7 (8) | 1 (2)
Neutropenic colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1)
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 2 (2)
Small intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 14 (16) | 2 (2)
Subileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 6 (6) | 8 (10)
Adverse drug reaction (General disorders) | 1 (2) | 0 (0)
Asthenia (General disorders) | 3 (11) | 4 (4)
Chest pain (General disorders) | 1 (1) | 2 (2)
Death (General disorders) | 5 (5) | 3 (3)
Disease progression (General disorders) | 1 (1) | 2 (2)
Fatigue (General disorders) | 12 (18) | 6 (6)
General physical health deterioration (General disorders) | 5 (6) | 1 (1)
Malaise (General disorders) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 2 (2) | 1 (1)
Multi-organ failure (General disorders) | 1 (1) | 1 (1)
Non-cardiac chest pain (General disorders) | 2 (2) | 3 (3)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 2 (2) | 2 (2)
Peripheral swelling (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 10 (10) | 10 (10)
Sudden death (General disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Jaundice (Hepatobiliary disorders) | 0 (0) | 1 (1)
Anaphylactic shock (Immune system disorders) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (2) | 2 (2)
Anal abscess (Infections and infestations) | 2 (4) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis perforated (Infections and infestations) | 1 (1) | 0 (0)
Biliary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 2 (2) | 6 (7)
Bronchitis moraxella (Infections and infestations) | 0 (0) | 1 (1)
Bronchopneumonia (Infections and infestations) | 1 (1) | 0 (0)
Candida infection (Infections and infestations) | 1 (1) | 0 (0)
Catheter site infection (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 3 (4) | 0 (0)
Cellulitis staphylococcal (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 2 (2) | 1 (1)
Device related infection (Infections and infestations) | 1 (1) | 2 (2)
Device related sepsis (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 3 (4) | 0 (0)
Empyema (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 2 (2) | 0 (0)
Lobar pneumonia (Infections and infestations) | 7 (7) | 8 (8)
Localised infection (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 2 (2) | 1 (3)
Lung infection (Infections and infestations) | 3 (6) | 5 (5)
Neutropenic infection (Infections and infestations) | 1 (1) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 2 (2) | 2 (2)
Oral candidiasis (Infections and infestations) | 2 (2) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 1 (1) | 0 (0)
Pelvic abscess (Infections and infestations) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 2 (2) | 0 (0)
Pharyngitis (Infections and infestations) | 3 (3) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 (0) | 3 (3)
Pneumonia (Infections and infestations) | 37 (43) | 41 (48)
Pneumonia bacterial (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia escherichia (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia pneumococcal (Infections and infestations) | 0 (0) | 2 (2)
Pneumonia staphylococcal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia streptococcal (Infections and infestations) | 1 (1) | 1 (1)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 3 (3) | 3 (3)
Sepsis (Infections and infestations) | 3 (3) | 2 (2)
Septic shock (Infections and infestations) | 2 (3) | 3 (3)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Stenotrophomonas sepsis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 4 (4)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Pubis fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Suture related complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic arthropathy (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1)
Diagnostic aspiration (Investigations) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1)
International normalised ratio increased (Investigations) | 0 (0) | 1 (1)
Liver function test abnormal (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 9 (10) | 3 (3)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 15 (17) | 15 (18)
Failure to thrive (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (3)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 4 (4) | 3 (3)
Hypovolaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Spinal disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intracranial tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 5 (6)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (4) | 3 (3)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (6) | 7 (10)
Pericardial effusion malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumour compression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 1 (1)
Brain oedema (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Cognitive disorder (Nervous system disorders) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 3 (3) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (2) | 2 (2)
Hemiparesis (Nervous system disorders) | 1 (2) | 0 (0)
Hemiplegia (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Ivth nerve paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 1 (2) | 0 (0)
Migraine with aura (Nervous system disorders) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Paraparesis (Nervous system disorders) | 1 (1) | 0 (0)
Peroneal nerve palsy (Nervous system disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Radicular syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Senile dementia (Nervous system disorders) | 1 (2) | 0 (0)
Stupor (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 4 (4) | 4 (4)
Toxic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 1 (2) | 0 (0)
Vocal cord paresis (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 7 (7) | 1 (1)
Conversion disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 1 (2)
Echolalia (Psychiatric disorders) | 0 (0) | 1 (1)
Mania (Psychiatric disorders) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1) | 1 (1)
Acute prerenal failure (Renal and urinary disorders) | 0 (0) | 1 (2)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 4 (8) | 2 (2)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 6 (6)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Catarrh (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 5 (7) | 4 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 (12) | 26 (32)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 7 (9) | 6 (7)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 9 (10) | 21 (23)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Pulmonary bulla (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 12 (13)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (5)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 9 (10)
Respiratory tract haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hospitalisation (Surgical and medical procedures) | 1 (1) | 0 (0)
Lung lobectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Aortic aneurysm rupture (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 2 (3) | 2 (2)
Hypertension (Vascular disorders) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 3 (3) | 4 (5)
Iliac artery occlusion (Vascular disorders) | 0 (0) | 1 (1)
Jugular vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1)
Peripheral artery aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Superior vena cava syndrome (Vascular disorders) | 0 (0) | 1 (1)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ramucirumab and Docetaxel (N=627) | Placebo and Docetaxel (N=618)
Anaemia (Blood and lymphatic system disorders) | 135 (306) | 174 (399)
Leukopenia (Blood and lymphatic system disorders) | 79 (259) | 68 (151)
Neutropenia (Blood and lymphatic system disorders) | 228 (547) | 188 (415)
Thrombocytopenia (Blood and lymphatic system disorders) | 51 (114) | 27 (48)
Lacrimation increased (Eye disorders) | 85 (100) | 29 (31)
Abdominal pain (Gastrointestinal disorders) | 56 (69) | 35 (41)
Constipation (Gastrointestinal disorders) | 107 (135) | 110 (132)
Diarrhoea (Gastrointestinal disorders) | 200 (338) | 175 (226)
Dyspepsia (Gastrointestinal disorders) | 37 (47) | 18 (25)
Nausea (Gastrointestinal disorders) | 170 (236) | 173 (256)
Stomatitis (Gastrointestinal disorders) | 143 (245) | 81 (104)
Vomiting (Gastrointestinal disorders) | 88 (117) | 86 (119)
Asthenia (General disorders) | 72 (178) | 65 (127)
Fatigue (General disorders) | 287 (623) | 260 (524)
Mucosal inflammation (General disorders) | 103 (167) | 43 (53)
Oedema peripheral (General disorders) | 107 (149) | 55 (86)
Pain (General disorders) | 35 (40) | 33 (37)
Pyrexia (General disorders) | 100 (148) | 79 (114)
Neutrophil count decreased (Investigations) | 112 (281) | 89 (193)
Platelet count decreased (Investigations) | 36 (104) | 9 (20)
Weight decreased (Investigations) | 67 (84) | 49 (56)
White blood cell count decreased (Investigations) | 58 (148) | 50 (219)
Decreased appetite (Metabolism and nutrition disorders) | 189 (290) | 163 (221)
Dehydration (Metabolism and nutrition disorders) | 39 (47) | 24 (31)
Hyperglycaemia (Metabolism and nutrition disorders) | 39 (83) | 25 (49)
Arthralgia (Musculoskeletal and connective tissue disorders) | 71 (110) | 51 (86)
Back pain (Musculoskeletal and connective tissue disorders) | 73 (113) | 56 (83)
Bone pain (Musculoskeletal and connective tissue disorders) | 31 (40) | 36 (57)
Myalgia (Musculoskeletal and connective tissue disorders) | 79 (123) | 65 (110)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 50 (60) | 26 (31)
Dizziness (Nervous system disorders) | 43 (54) | 46 (52)
Dysgeusia (Nervous system disorders) | 69 (83) | 46 (55)
Headache (Nervous system disorders) | 66 (88) | 65 (78)
Paraesthesia (Nervous system disorders) | 38 (49) | 36 (46)
Peripheral sensory neuropathy (Nervous system disorders) | 74 (121) | 60 (102)
Insomnia (Psychiatric disorders) | 69 (78) | 54 (55)
Cough (Respiratory, thoracic and mediastinal disorders) | 137 (194) | 131 (169)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 38 (49) | 23 (23)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 150 (220) | 148 (207)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 116 (149) | 41 (45)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 36 (38) | 31 (37)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 49 (65) | 30 (39)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 40 (61) | 34 (41)
Alopecia (Skin and subcutaneous tissue disorders) | 163 (192) | 156 (176)
Nail discolouration (Skin and subcutaneous tissue disorders) | 41 (45) | 27 (27)
Rash (Skin and subcutaneous tissue disorders) | 44 (56) | 36 (51)
Hypertension (Vascular disorders) | 67 (129) | 29 (107)

LIMITATIONS AND CAVEATS:
Three participants randomized to placebo and docetaxel received 1 dose of ramucirumab in error. They are included in the placebo and docetaxel arm in the ITT population and are included in the ramucirumab and docetaxel arm in the Safety population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators agreed to delay independently publishing or disclosing data, findings or conclusions from the study except as part of a multi-center publication. Upon study publication or if the draft publication is not produced within approximately 6 months of the final report of the study results, investigators may independently publish, subject to confidential information review/redaction by sponsor. The sponsor may request publication delay up to 90 days to seek patent protection.